CLINICAL TRIAL: NCT07099859
Title: Effect of Losartan on the Neurohumoral Axis and Ventricular Remodeling of Patients With Severe Aortic Regurgitation Undergoing Valve Surgery
Acronym: ARBNP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vitor Emer Egypto Rosa (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor-Investigator, Vitor Emer Egypto Rosa, Principal investigator, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 81900224.0.0000.0068; 2023/15710-5 (Other: FAPESP)
Record Dates: First submitted 2025-07-08; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Heart Valve Diseases; Left Ventricle Remodeling; Aortic Regurgitation Disease; Heart Failure Congestive; Natriuretic Peptide, Brain
Keywords: aortic regurgitation; valve disease; heart surgery; heart failure; losartan; Brain natriuretic peptide - BNP; biomarkers; renin-angiotensin-aldosterone system; neurohumoral axis
MeSH Terms: conditions — Heart Valve Diseases; Ventricular Remodeling; Heart Failure; Aortic Valve Insufficiency | interventions — Losartan

STUDY DESIGN:
Intervention Model Description: This is a pilot, randomized, double-blind clinical study with a sample of 60 patients, who will be randomized in a 1:1 ratio. Patients in both arms will be assessed at 4 time points: randomization, 1, 3 and 12 months after surgery, undergoing a 6-minute walk test and Short-Form Health Survey (SF-36v2) quality of life questionnaire, laboratory tests including NT-proBNP, electrolytes and renal function, as well as a complete echocardiographic evaluation.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losartan group (Experimental): losartan 50 mg/day
  Interventions: Drug: Losartan 50 mg
- placebo group (Placebo Comparator): placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan 50 mg — Losartan 50 mg per day
  Arms: Losartan group
Drug: Placebo — Placebo 1 pill per day
  Arms: placebo group

SUMMARY:
Why Is This Study Important? The heart has valves that help control blood flow. Aortic regurgitation (AR) is a condition where one of these valves (the aortic valve) doesn't close properly, causing blood to leak back into the heart. Over time, this makes the heart work harder and grow larger (remodeling) to keep up. Many patients with severe AR need valve replacement surgery to fix this problem.

After surgery, the heart doesn't have to work as hard, and over time, it can shrink back to a healthier size (reverse remodeling). However, doctors don't know if medications can help speed up or improve this healing process. This study aims to find out if a common blood pressure medication, losartan, can help the heart recover better after surgery.

What Do the Investigators Already Know? Doctors often prescribe medications like ACE inhibitors, angiotensin receptor blockers (ARBs), beta-blockers, and spironolactone to people with heart failure because these drugs help the heart function better and prevent worsening disease. However, these medications haven't been studied in people with valve disease because most major research studies excluded patients with valve problems.

Even though there is not strong evidence, many doctors prescribe these medications after valve surgery, assuming they might be helpful. But is that really the case? That's the question this study hopes to answer.

What Is This Study About?

This study will test whether losartan, a medication often used for high blood pressure, can help hearts recover better after aortic valve replacement surgery. The researchers will compare two groups of patients:

* One group will take losartan (50 mg per day) after surgery.
* The other group will take a placebo (a pill with no active medication).

By comparing these two groups, the study will determine whether losartan helps the heart shrink back to a normal size faster and function better after surgery.

How Will the Study Work? Who? 60 patients with severe AR who are having aortic valve replacement surgery.

How? Patients will be randomly placed into one of the two groups (losartan or placebo).

For how long? Patients will be followed for one year after surgery. What Will Be Measured?

Doctors will check patients four times: before surgery, and 1 month, 3 months, and 12 months after surgery. At each visit, the investigators will measure:

* NT-proBNP levels: A blood test that tells us how much strain the heart is under. Lower levels mean the heart is recovering well.
* Echocardiogram: An ultrasound of the heart to check its size and function.
* 6-minute walk test: To see if patients feel stronger and can exercise better.
* Quality of life survey: To understand how patients feel physically and emotionally.
* Kidney function and electrolyte levels: To check for medication side effects.

Why Is This Study Exciting? This is the first study to test whether a medication can help the heart heal better after valve surgery. If losartan proves beneficial, it could change how doctors treat patients after surgery and lead to better recovery, stronger hearts, and healthier lives.

Many people with aortic regurgitation have to wait until their symptoms get worse before patients can have surgery. If this study finds that medication can speed up healing, it could help doctors treat valve disease more effectively and improve long-term outcomes for patients.

What Happens Next? If losartan is found to be helpful, this study could lead to larger research trials and, eventually, new treatment guidelines for people who have had aortic valve surgery. If it doesn't help, doctors will know not to prescribe it unnecessarily, preventing unnecessary side effects and costs for patients. Either way, the results will help improve care for people with heart valve disease.

By participating in this study, patients are helping researchers discover new ways to improve heart health and recovery after surgery.

DETAILED DESCRIPTION:
Pharmacological therapy targeting the neurohumoral axis have emerged as the cornerstone of Heart Failure (HF) treatment. The angiotensin-converting enzyme inhibitors, angiotensin receptor blockers (ARBs), spironolactone, beta-blockers and neprilysin inhibitors act on the neurohumoral axis, having prognostic impact with proven benefits in terms of ventricular remodeling, morbidity and mortality. However, these drugs have not been tested in the context of valvular cardiomyopathy, as pivotal studies excluded patients with valve disease. There are robust evidences that medical treatment does not reduce mortality in the preoperative phase of valve disease, acting only on symptom management. However, in the period after valve surgery, there is absence of data regarding benefit of medical therapy focused on the neurohumoral axis. Aortic regurgitation represents a condition characterized by pronounced ventricular remodeling during the asymptomatic phase, often developing significant reverse remodeling after surgery. Consequently, it presents as a very interesting model for studying the impact of renin-angiotensin-aldosterone system inhibition after valve intervention. Currently, clinicians frequently precribe drugs targeting the neurohumoral axis in the postoperative phase for these patients, extrapolating from findings in classical HF studies. However, there is no evidence in the literature for this approach, which is common in clinical practice. Therefore, this study aims to assess the impact of the use of the ARB losartan on neurohumoral remodeling in the postoperative period of patients with aortic regurgitation undergoing valve surgery, measuring NT-proBNP, a natriuretic peptide strongly associated with ventricular remodeling. The primary objective of the study is to compare NT-proBNP values in patients taking losartan 50 mg/day versus placebo in the first 3 months after aortic valve replacement for severe aortic regurgitation. This is a pilot, randomized, double-blind clinical study with a sample of 60 patients, who will be randomized in a 1:1 ratio. Patients in both arms will be assessed at 4 time points: randomization, 1, 3 and 12 months after surgery, undergoing a 6-minute walk test and Short-Form Health Survey (SF-36v2) quality of life questionnaire, laboratory tests including NT-proBNP, electrolytes and renal function, as well as a complete echocardiographic evaluation.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years;
* Postoperative period of aortic valve replacement surgery due to severe aortic regurgitation of any etiology;
* Signed Informed Consent Form.

Exclusion Criteria:

To avoid potential bias in data interpretation, the following patients will be excluded:

* Those who underwent cardiac surgery in the context of cardiogenic shock or infective endocarditis;
* Patients with ischemic cardiomyopathy;
* Patients with other significant concomitant valvular diseases.

Patients with conditions where losartan use may be harmful will also be excluded, including:

* Chronic kidney disease with an estimated glomerular filtration rate (eGFR < 30 ml/min/1.73 m²);
* Systolic blood pressure (SBP) < 90 mmHg at the time of randomization;
* Elevated serum potassium (K > 5.5 mEq/L) at the time of randomization;
* Pregnancy;
* Known intolerance or allergy to losartan.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Change of NT-proBNP during the first 3 months after aortic valve surgery in patients with severe aortic regurgitation. | 3 months
  The primary outcome of the study will be to evaluate the reduction of NT-proBNP during the first 3 months after aortic valve surgery in patients with severe aortic regurgitation.

SECONDARY OUTCOMES:
Evaluation of the effects of losartan on NT-proBNP levels after aortic valve surgery in 1 and 12 months. | 12 months
  -NT-proBNP (pg/ml) reduction at 1 and 12 months, compared to pre-discharge values.
Evaluation of the effects of losartan on cardiac remodeling after aortic valve surgery in 1, 3 and 12 months. | 1, 3, and 12 months
  -Left ventricular reverse remodeling: ejection fraction (%) at 1, 3, and 12 months.
Evaluation of the effects of losartan on quality of life after aortic valve surgery in 1, 3 and 12 months. | 1, 3 and 12 months
  -Quality of life questionnare: Short-Form Health Survey (SF-36v2) with values ranging from 0 to 100 points (100 = best possible health status) at 1, 3, and 12 months.
Evaluation of the effects of losartan on functional capacity after aortic valve surgery in 1, 3 and 12 months | 1, 3 and 12 months
  - 6-minute walk test (meters) at 1, 3, and 12 months.
Evaluation of the effects of losartan on kidney function after aortic valve surgery in 1, 3 and 12 months. | 1, 3 and 12 months
  -Acute kidney injury (KDIGO criteria) at 1, 3, and 12 months: Stage 1: 1.5-1.9× baseline or ≥0.3 mg/dL increase Stage 2: 2.0-2.9× baseline Stage 3: 3× baseline, ≥4.0 mg/dL increase, dialysis, or clearance <35ml/min/1.73m² -Hyperkalemia (K > 5.6 mEq/L)
Evaluation of the effects of losartan on major cardiovascular events after aortic valve surgery in 1, 3 and 12 months. | 1, 3 and 12 months
  * Rate of cardiac rehospitalization, cardiovascular and all-cause mortality
  * Rate of MACE: myocardial infarction, stroke, or cardiovascular death.
Evaluation of the effects of losartan on cardiac remodeling after aortic valve surgery in 1, 3 and 12 months. | 1, 3, and 12 months
  -Left ventricular reverse remodeling: left ventricular mass index (g/m2) at 1, 3, and 12 months.
Evaluation of the effects of losartan on cardiac remodeling after aortic valve surgery in 1, 3 and 12 months. | 1, 3, and 12 months
  -Left ventricular reverse remodeling: left ventricular diameters (mm) at 1, 3, and 12 months.
Evaluation of the effects of losartan on cardiac remodeling after aortic valve surgery in 1, 3 and 12 months. | 1, 3, and 12 months
  -Left ventricular reverse remodeling: left ventricular volumes (ml) at 1, 3, and 12 months.
Evaluation of the effects of losartan on cardiac remodeling after aortic valve surgery in 1, 3 and 12 months. | 1, 3, and 12 months
  -Left ventricular reverse remodeling: left ventricular global longitudinal strain (%) at 1, 3, and 12 months.
Evaluation of the effects of losartan on cardiac remodeling after aortic valve surgery in 1, 3 and 12 months. | 1, 3, and 12 months
  -Left ventricular reverse remodeling: left ventricular myocardial work (GWI: global left ventricular myocardial work index-mmHg%) at 1, 3, and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Vitor E. E. Rosa, MD, PhD, Principal Investigator — Heart Institute of the School of Medicine of the University of São Paulo
Locations (1):
- Heart Institute of the School of Medicine of the University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Eichhorn EJ, Bristow MR. Medical therapy can improve the biological properties of the chronically failing heart. A new era in the treatment of heart failure. Circulation. 1996 Nov 1;94(9):2285-96. doi: 10.1161/01.cir.94.9.2285. PMID 8901684
- [Background] Lang CC, Struthers AD. Targeting the renin-angiotensin-aldosterone system in heart failure. Nat Rev Cardiol. 2013 Mar;10(3):125-34. doi: 10.1038/nrcardio.2012.196. Epub 2013 Jan 15. PMID 23319100
- [Background] Cohn JN, Tognoni G; Valsartan Heart Failure Trial Investigators. A randomized trial of the angiotensin-receptor blocker valsartan in chronic heart failure. N Engl J Med. 2001 Dec 6;345(23):1667-75. doi: 10.1056/NEJMoa010713. PMID 11759645
- [Background] Wong M, Staszewsky L, Latini R, Barlera S, Volpi A, Chiang YT, Benza RL, Gottlieb SO, Kleemann TD, Rosconi F, Vandervoort PM, Cohn JN; Val-HeFT Heart Failure Trial Investigators. Valsartan benefits left ventricular structure and function in heart failure: Val-HeFT echocardiographic study. J Am Coll Cardiol. 2002 Sep 4;40(5):970-5. doi: 10.1016/s0735-1097(02)02063-6. PMID 12225725
- [Background] Young JB, Dunlap ME, Pfeffer MA, Probstfield JL, Cohen-Solal A, Dietz R, Granger CB, Hradec J, Kuch J, McKelvie RS, McMurray JJ, Michelson EL, Olofsson B, Ostergren J, Held P, Solomon SD, Yusuf S, Swedberg K; Candesartan in Heart failure Assessment of Reduction in Mortality and morbidity (CHARM) Investigators and Committees. Mortality and morbidity reduction with Candesartan in patients with chronic heart failure and left ventricular systolic dysfunction: results of the CHARM low-left ventricular ejection fraction trials. Circulation. 2004 Oct 26;110(17):2618-26. doi: 10.1161/01.CIR.0000146819.43235.A9. Epub 2004 Oct 18. PMID 15492298
- [Background] Pfeffer MA, Swedberg K, Granger CB, Held P, McMurray JJ, Michelson EL, Olofsson B, Ostergren J, Yusuf S, Pocock S; CHARM Investigators and Committees. Effects of candesartan on mortality and morbidity in patients with chronic heart failure: the CHARM-Overall programme. Lancet. 2003 Sep 6;362(9386):759-66. doi: 10.1016/s0140-6736(03)14282-1. PMID 13678868
- [Background] Della Corte A, Salerno G, Chiosi E, Iarussi D, Santarpino G, Miraglia M, Naviglio S, De Feo M. Preoperative, postoperative and 1-year follow-up N-terminal pro-B-type natriuretic peptide levels in severe chronic aortic regurgitation: correlations with echocardiographic findings. Interact Cardiovasc Thorac Surg. 2008 May;7(3):419-24; discussion 424. doi: 10.1510/icvts.2007.168039. Epub 2008 Mar 19. PMID 18353850
- [Background] Song BG, Park YH, Kang GH, Chun WJ, Oh JH, Choi JO, Lee SC, Park SW, Oh JK, Sung KI, Park P, Jeon ES. Preoperative, postoperative and one-year follow-up of N-terminal pro-B-type natriuretic peptide levels in volume overload of aortic regurgitation: comparison with pressure overload of aortic stenosis. Cardiology. 2010;116(4):286-91. doi: 10.1159/000318019. Epub 2010 Sep 22. PMID 20861629
- [Background] Rodriguez-Gabella T, Catala P, Munoz-Garcia AJ, Nombela-Franco L, Del Valle R, Gutierrez E, Regueiro A, Jimenez-Diaz VA, Ribeiro HB, Rivero F, Fernandez-Diaz JA, Pibarot P, Alonso-Briales JH, Tirado-Conte G, Moris C, Diez Del Hoyo F, Jimenez-Britez G, Zaderenko N, Alfonso F, Gomez I, Carrasco-Moraleja M, Rodes-Cabau J, San Roman Calvar JA, Amat-Santos IJ. Renin-Angiotensin System Inhibition Following Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2019 Aug 6;74(5):631-641. doi: 10.1016/j.jacc.2019.05.055. PMID 31370954
- [Background] Symeonides P, Koulouris S, Vratsista E, Triantafyllou K, Ioannidis G, Thalassinos N, Katritsis D. Both ramipril and telmisartan reverse indices of early diabetic cardiomyopathy: a comparative study. Eur J Echocardiogr. 2007 Dec;8(6):480-6. doi: 10.1016/j.euje.2006.09.005. Epub 2006 Nov 17. PMID 17113349
- [Background] Weber M, Arnold R, Rau M, Elsaesser A, Brandt R, Mitrovic V, Hamm C. Relation of N-terminal pro B-type natriuretic peptide to progression of aortic valve disease. Eur Heart J. 2005 May;26(10):1023-30. doi: 10.1093/eurheartj/ehi236. Epub 2005 Mar 21. PMID 15781428
- [Background] Tarasoutchi F, Grinberg M, Spina GS, Sampaio RO, Cardoso Lu, Rossi EG, Pomerantzeff P, Laurindo F, da Luz PL, Ramires JA. Ten-year clinical laboratory follow-up after application of a symptom-based therapeutic strategy to patients with severe chronic aortic regurgitation of predominant rheumatic etiology. J Am Coll Cardiol. 2003 Apr 16;41(8):1316-24. doi: 10.1016/s0735-1097(03)00129-3. PMID 12706927
- [Background] Weiner RB, Baggish AL, Chen-Tournoux A, Marshall JE, Gaggin HK, Bhardwaj A, Mohammed AA, Rehman SU, Barajas L, Barajas J, Gregory SA, Moore SA, Semigran MJ, Januzzi JL Jr. Improvement in structural and functional echocardiographic parameters during chronic heart failure therapy guided by natriuretic peptides: mechanistic insights from the ProBNP Outpatient Tailored Chronic Heart Failure (PROTECT) study. Eur J Heart Fail. 2013 Mar;15(3):342-51. doi: 10.1093/eurjhf/hfs180. Epub 2012 Nov 6. PMID 23132825
- [Background] Daubert MA, Adams K, Yow E, Barnhart HX, Douglas PS, Rimmer S, Norris C, Cooper L, Leifer E, Desvigne-Nickens P, Anstrom K, Fiuzat M, Ezekowitz J, Mark DB, O'Connor CM, Januzzi J, Felker GM. NT-proBNP Goal Achievement Is Associated With Significant Reverse Remodeling and Improved Clinical Outcomes in HFrEF. JACC Heart Fail. 2019 Feb;7(2):158-168. doi: 10.1016/j.jchf.2018.10.014. Epub 2019 Jan 2. PMID 30611722
- [Background] Pitt B, Poole-Wilson PA, Segal R, Martinez FA, Dickstein K, Camm AJ, Konstam MA, Riegger G, Klinger GH, Neaton J, Sharma D, Thiyagarajan B. Effect of losartan compared with captopril on mortality in patients with symptomatic heart failure: randomised trial--the Losartan Heart Failure Survival Study ELITE II. Lancet. 2000 May 6;355(9215):1582-7. doi: 10.1016/s0140-6736(00)02213-3. PMID 10821361
- [Background] Oremus M, McKelvie R, Don-Wauchope A, Santaguida PL, Ali U, Balion C, Hill S, Booth R, Brown JA, Bustamam A, Sohel N, Raina P. A systematic review of BNP and NT-proBNP in the management of heart failure: overview and methods. Heart Fail Rev. 2014 Aug;19(4):413-9. doi: 10.1007/s10741-014-9440-0. PMID 24953975